CLINICAL TRIAL: NCT01251601
Title: The Effect of Pregnancy on the Pharmacokinetics of Isentress®: A Longitudinal Investigation in the Second and Third Trimesters
Brief Title: The Effect of Pregnancy on the PK of Isentress®: A Longitudinal Investigation in the Second and Third Trimesters
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn due to inability to recruit eligible participants
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-1691
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2012-01

CONDITIONS: HIV; Pregnancy
MeSH Terms: interventions — Pharmacokinetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Raltegravir in Pregnancy: HIV positive pregnant women currently on raltegravir as part of combination antiretroviral therapy
  Interventions: Other: Pharmacokinetics

INTERVENTIONS:
Other: Pharmacokinetics — Up to three 12 hour PK sampling sessions, one in the second trimester, one in the third trimester and one post partum

SUMMARY:
The purpose of this study is to determine whether pregnancy affects the blood concentrations of raltegravir by comparing the second trimester and third trimester drug concentrations with post partum.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infected
* Pregnant
* At least 18 years of age
* Planning to initiate or currently received raltegravir as part of an antiretroviral regimen with plans to continue at least 8-10 weeks post partum

Exclusion Criteria:

* Less than 18 years of age
* Hemoglobin <9 g/dL or Hematocrit <27.3 at screening

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by their HIV clinic providers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — UNC Chapel Hill; Kristine B Patterson, MD, Principal Investigator — UNC Chapel Hill